CLINICAL TRIAL: NCT02723916
Title: Parent Training in Pediatric Care: A Self Directed Tablet-Based Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Susie Breitenstein, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ORA# 15012705
Record Dates: First submitted 2016-01-21; First posted 2016-03-31 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Parent Training; Primary Care
Keywords: Parents; Child; Preschool; eHealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: ezParent Program (Experimental)
  Interventions: Behavioral: ezParent Program
- Control: Health-e Kids App (Active Comparator)
  Interventions: Behavioral: Health-e Kids Control App

INTERVENTIONS:
Behavioral: ezParent Program — Tablet-based behavioral parent training program.
  Other Names: previously called eCPP
  Arms: Intervention: ezParent Program
Behavioral: Health-e Kids Control App — Tablet based health promotion information App
  Arms: Control: Health-e Kids App

SUMMARY:
High quality and effective parenting in the preschool years is connected with long term positive child behavior and mental health outcomes. The purpose of the study, "Parent Training in Pediatric Primary Care: A Self-directed Tablet-based Approach," is to test the outcomes and implementation of a tablet-based parent training program in Pediatric Primary Care. Testing and evaluating the implementation of digitally delivered programs is important to increase the ease, reach, sustainability, and integration of mental health prevention into primary care settings.

DETAILED DESCRIPTION:
One in four young children in the United States faces poverty-associated risks that make her or him more likely to have mental health and behavior problems. These problems, left untreated, can have long-term social, emotional, and behavioral consequences. High-quality parenting in the preschool years can substantially buffer the negative effects of socioeconomic adversity on children's mental health and behavior. However, most parent training programs use face-to-face delivery models resulting in barriers to participation and limited reach to those most in need. Testing the efficacy and implementation of alternative delivery models is needed to (a) increase the reach and sustainability of parent training interventions and (b) address the barriers to parent participation and implementation of such programs, specifically in primary health care settings. The parent training program proposed in this study is a digital adaptation (tablet-based) of the evidence-based based Chicago Parent Program (CPP) called the ezParent Program. The purpose of this study is to evaluate the efficacy, cost-effectiveness, and implementation process of delivering the ezParent in pediatric primary care sites serving low-income, urban families. The specific aims of the study are: (1) Test the direct effects of the 6-module ezParent Program on parenting outcomes (parenting behavior, parenting self-efficacy, and parenting stress) and child outcomes (child problem and prosocial behavior) compared to an enhanced usual care control condition among low-income parents with young children seen in primary care settings; (2) Compare the cost-effectiveness of the ezParent intervention relative to the control condition for the parenting and child outcomes; and (3) Quantify the levels of program implementation of the ezParent Program in primary care using the RE-AIM framework. The efficacy of the ezParent Program will be tested using a randomized clinical trial design with 312 parents of 2- to 5-year-old children from pediatric primary care settings. Data on parenting and child behavior outcomes will be obtained from all participants at baseline, and 3, 6, and 12 months post baseline. A descriptive design guided by the RE-AIM framework and cost-effectiveness analysis will evaluate the implementation of the ezParent Program in the pediatric primary care sites.

Integrating and evaluating the implementation of the ezParent Program is an innovative opportunity to promote parenting with potential for universal access to the preschool (2- to 5-year-olds) population and potential for low cost by building on existing infrastructure. Findings from this study will lay the foundation for full-scale implementation of the ezParent Program in pediatric primary care settings and subsequent implementation and dissemination research.

ELIGIBILITY:
Inclusion Criteria:

* parent, legal guardian, or primary caregiver for the target child,
* target child is 2-5 years old,
* child receives care at the primary practice implementation site,
* parent can speak and read English.

Exclusion Criteria:

* Only one parent per family
* Parent does not meet inclusion criteria.
* Parent previously used the ezPARENT program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breitenstein SM, Schoeny M, Risser H, Johnson T. A study protocol testing the implementation, efficacy, and cost effectiveness of the ezParent program in pediatric primary care. Contemp Clin Trials. 2016 Sep;50:229-37. doi: 10.1016/j.cct.2016.08.017. Epub 2016 Aug 31. PMID 27592122
- [Result] Breitenstein SM, Laurent S, Pabalan L, Risser HJ, Roper P, Saba MT, Schoeny M. Implementation findings from an effectiveness-implementation trial of tablet-based parent training in pediatric primary care. Fam Syst Health. 2019 Dec;37(4):282-290. doi: 10.1037/fsh0000447. Epub 2019 Oct 17. PMID 31621349
- [Result] Fehrenbacher C, Schoeny ME, Reed M, Shattell M, Breitenstein SM. Referral to Digital Parent Training in Primary Care: Facilitators and Barriers. Clin Pract Pediatr Psychol. 2020 Sep;8(3):268-277. doi: 10.1037/cpp0000367. PMID 35821979
- [Derived] Breitenstein SM, Fehrenbacher C, Holod AF, Schoeny ME. A Randomized Trial of Digitally Delivered, Self-Administered Parent Training in Primary Care: Effects on Parenting and Child Behavior. J Pediatr. 2021 Apr;231:207-214.e4. doi: 10.1016/j.jpeds.2020.12.016. Epub 2020 Dec 16. PMID 33338496

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from April 2016 - April 2018
Pre-assignment Details: No pre-assignment in study.
Period: Overall Study
Arm/Group | Intervention: ezParent Program | Control: Health-e Kids App
Started | 144 | 143
Completed | 135 | 137
Not Completed | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention: ezParent Program | Control: Health-e Kids App | Total
Number analyzed (Participants) | 144 | 143 | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (8.16) | 32.9 (7.70) | 32.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 136 | 272
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 43 | 77
  Not Hispanic or Latino | 110 | 100 | 210
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 99 | 75 | 174
  White | 17 | 24 | 41
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 21 | 31 | 52
Region of Enrollment [Number; unit: participants]
  United States | 144 | 143 | 287

OUTCOME MEASURES:

1. Primary Outcome: Parenting Behaviors
Description: Measured by the Parent Questionnaire (PQ)
  Scale scores reported:
  Warmth (scale range 1-5) - higher score indicates improvement Parent Follow Through (scale range 1-5) - higher score indicates improvement Corporal punishment (scale range 1-5) - lower score indicates improvement
Time Frame: T1 = baseline; T2 = 3-months post baseline; T3 = 6-months post baseline; T4 = 12-months post baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: ezParent Program | Control: Health-e Kids App
Number analyzed (Participants) | 144 | 143
score on a scale
  Parental Warmth (T1) | 4.30 (0.46) | 4.27 (0.41)
  Parental Warmth (T2) | 4.26 (0.42) | 4.25 (.41)
  Parental Warmth (T3) | 4.29 (.39) | 4.3 (.44)
  Parental Warmth (T4) | 4.27 (.46) | 4.34 (.4)
  Parental Follow Through (T1) | 3.46 (0.68) | 3.37 (0.78)
  Parental Follow Through (T2) | 3.47 (0.75) | 3.49 (.71)
  Parental Follow Through (T3) | 3.58 (.77) | 3.52 (.7)
  Parental Follow Through (T4) | 3.64 (.75) | 3.59 (.76)
  Corporal Punishment (T1) | 1.43 (0.49) | 1.51 (0.53)
  Corporal Punishment (T2) | 1.47 (0.55) | 1.49 (0.55)
  Corporal Punishment (T3) | 1.44 (.59) | 1.47 (.57)
  Corporal Punishment (T4) | 1.42 (.58) | 1.39 (.5)

2. Secondary Outcome: Change in Parent Behaviors
Description: Measured by the Parenting Young Children (PARYC) Reporting scales (scale range 1-7) (higher scores indicate more effective/improved parenting) Supporting good behavior Setting limits Proactive parenting
Time Frame: T1 = baseline; T2 = 3-months post baseline; T3 = 6-months post baseline; T4 = 12-months post baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: ezParent Program | Control: Health-e Kids App
Number analyzed (Participants) | 144 | 143
score on a scale
  Supporting Good Behavior (T1) | 5.63 (0.96) | 5.70 (0.98)
  Supporting Good Behavior (T2) | 5.36 (1.11) | 5.65 (1.00)
  Supporting Good Behavior (T3) | 5.54 (.99) | 5.7 (1.07)
  Supporting Good Behavior (T4) | 5.53 (1.15) | 5.85 (.87)
  Setting Limits (T1) | 5.17 (1.18) | 5.24 (1.04)
  Setting Limits (T2) | 5.14 (1.10) | 5.23 (1.06)
  Setting Limits (T3) | 5.31 (1.07) | 5.37 (1.19)
  Setting Limits (T4) | 5.41 (1.10) | 5.52 (1.12)
  Proactive Parenting (T1) | 5.08 (1.32) | 5.13 (1.27)
  Proactive Parenting (T2) | 5.04 (1.12) | 5.08 (1.26)
  Proactive Parenting (T3) | 5.2 (1.26) | 5.3 (1.21)
  Proactive Parenting (T4) | 5.29 (1.27) | 5.48 (1.28)

3. Secondary Outcome: Change in Child Behavior Problems
Description: Strengths and Difficulties Questionnaire (SDQ) scales (range 0-10) Emotional symptoms (higher scores indicate more difficulties) Conduct problems (higher scores indicate more difficulties) Hyperactivity/inattention (higher scores indicate more difficulties) Peer relationship problems (higher scores indicate more difficulties) Prosocial behavior (higher scores indicate more strengths)
Time Frame: T1 = baseline; T2 = 3-months post baseline; T3 = 6-months post baseline; T4 = 12-months post baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: ezParent Program | Control: Health-e Kids App
Number analyzed (Participants) | 144 | 143
score on a scale
  Emotion (T1) | 1.06 (1.39) | 1.12 (1.33)
  Emotion (T2) | 1.1 (1.61) | 1.03 (1.21)
  Emotion (T3) | 1.02 (1.43) | .97 (1.36)
  Emotion (T4) | 1.03 (1.44) | .92 (1.23)
  Conduct (T1) | 1.93 (1.90) | 1.94 (1.77)
  Conduct (T2) | 1.63 (1.79) | 1.77 (1.64)
  Conduct (T3) | 1.56 (1.83) | 1.75 (1.76)
  Conduct (T4) | 1.4 (1.81) | 1.53 (1.52)
  Hyper (T1) | 3.50 (2.29) | 3.38 (2.28)
  Hyper (T2) | 3.18 (2.26) | 3.46 (2.22)
  Hyper (T3) | 3.09 (2.49) | 2.91 (2.14)
  Hyper (T4) | 3.09 (2.32) | 2.84 (2.2)
  Peer (T1) | 1.62 (1.56) | 1.52 (1.64)
  Peer (T2) | 1.4 (1.6) | 1.53 (1.56)
  Peer (T3) | 1.27 (1.41) | 1.31 (1.47)
  Peer (T4) | 1.49 (1.71) | 1.45 (1.57)
  Prosocial (T1) | 8.01 (1.94) | 8.26 (1.74)
  Prosocial (T2) | 8.43 (1.94) | 8.24 (1.96)
  Prosocial (T3 | 8.5 (1.81) | 8.6 (1.55)
  Prosocial (T4) | 8.72 (1.92) | 8.45 (1.86)

4. Secondary Outcome: Change in Child Externalizing Behavior Problems
Description: Eyberg Child Behavior Inventory (ECBI) Problem scale (range 0-1) higher scores more problems Intensity scale (range 1-7) higher scores more intense problems
Time Frame: T1 = baseline; T2 = 3-months post baseline; T3 = 6-months post baseline; T4 = 12-months post baseline.
Population: Severity (intensity scale) 1 = never happens to 7 = always happening (higher scores more intense problems) - range is 1-7 Frequency (problem Scale of child behaviors. 0 = no; 1 = yes (higher scores more problems) Range 0-1
  T1 = baseline; T2 = 3-months post baseline; T3 = 6-months post baseline; T4 = 12-months post baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: ezParent Program | Control: Health-e Kids App
Number analyzed (Participants) | 144 | 143
score on a scale
  Problem Scale (T1) | 0.18 (0.22) | 0.19 (0.21)
  Problem Scale (T2) | .14 (.18) | .16 (.19)
  Problem Scale (T3) | .14 (.2) | .15 (.19)
  Problem Scale (T4) | .12 (.18) | .13 (.19)
  Intensity Scale (T1) | 2.80 (0.84) | 2.84 (0.80)
  Intensity Scale (T2) | 2.69 (.85) | 2.69 (.72)
  Intensity Scale (T3) | 2.64 (.8) | 2.67 (.75)
  Intensity Scale (T4) | 2.64 (.74) | 2.56 (.74)

5. Secondary Outcome: Change in Parenting Stress
Description: Parenting Stress Index-Short Form (PSI-SF) Scales (range 12-60): Higher scores indicate higher stress Parental distress Parent-child dysfunctional interaction Difficult child
Time Frame: T1 = baseline; T2 = 3-months post baseline; T3 = 6-months post baseline; T4 = 12-months post baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: ezParent Program | Control: Health-e Kids App
Number analyzed (Participants) | 144 | 143
score on a scale
  Parent Domain (T1) | 26.06 (9.58) | 25.53 (7.86)
  Parent Domain (T2) | 25.9 (9.26) | 25.25 (8.17)
  Parent Domain (T3) | 25.39 (10.04) | 25.41 (9.56)
  Parent Domain (T4) | 25.3 (9.72) | 24.64 (8.18)
  Parent-Child Domain (T1) | 20.28 (6.38) | 19.76 (6.05)
  Parent-Child Domain (T2) | 19.62 (6.5) | 20.02 (5.79)
  Parent-Child Domain (T3) | 19.62 (6.53) | 19.7 (6.87)
  Parent-Child Domain (T4) | 19.52 (6.03) | 19.62 (6.07)
  Child Domain (T1) | 24.72 (8.02) | 24.24 (6.86)
  Child Domain (T2) | 23.97 (7.62) | 24.34 (7.29)
  Child Domain (T3) | 23.37 (7.45) | 23.46 (7.66)
  Child Domain (T4) | 23.11 (7.18) | 23.18 (7.6)

6. Secondary Outcome: Change in Parenting Self-efficacy
Description: Parenting Sense of Competence Scale (PSOC) - Total Scale (Range 17-102) Higher scores indicate higher self efficacy
Time Frame: T1 = baseline; T2 = 3-months post baseline; T3 = 6-months post baseline; T4 = 12-months post baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: ezParent Program | Control: Health-e Kids App
Number analyzed (Participants) | 144 | 143
score on a scale
  Total Score (T1) | 71.07 (11.41) | 71.28 (10.62)
  Total Score (T2) | 71.51 (11.20) | 70.94 (10.7)
  Total Score (T3) | 72.99 (11.16) | 71.73 (12.24)
  Total Score (T4) | 72.9 (12.10) | 72.1 (11.00)

ADVERSE EVENTS:
Time Frame: 1 year
Description: No difference with definitions of adverse events and/or serious adverse events.
Arm/Group | Intervention: ezParent Program | Control: Health-e Kids App
All-Cause Mortality (participants affected / at risk) | 0/144 | 0/143
Serious Adverse Events (participants affected / at risk) | 0/144 | 0/143
Other Adverse Events (participants affected / at risk) | 0/144 | 0/143

LIMITATIONS AND CAVEATS:
No specific limitations related to the conduct of the study to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT02723916/Prot_SAP_000.pdf